CLINICAL TRIAL: NCT05586178
Title: Information Provision and Consistency Framing to Increase COVID-19 Booster Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey T. Fujimoto, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: covidbooster2
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; Vaccines
Keywords: COVID19; Vaccines; Text-messages; Patient Outreach; Behavioral Science; Information provision
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Holdout (No Intervention)
- Simple reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action
- Consistency reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action; Behavioral: Consistency framing
- Uniqueness information reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action; Behavioral: Information provision about the uniqueness of the bivalent booster
- Eligibility information reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action; Behavioral: Information provision about bivalent booster eligibility
- Severity information reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action; Behavioral: Information provision about the severity of COVID-19 symptoms
- Consistency and uniqueness information reminder (Experimental)
  Interventions: Behavioral: Reminder that facilitates action; Behavioral: Consistency framing; Behavioral: Information provision about the uniqueness of the bivalent booster

INTERVENTIONS:
Behavioral: Reminder that facilitates action — Patients will receive a text message reminding them that they can now get the bivalent COVID-19 booster and facilitating action. The message will contain a link to schedule a booster appointment at UCLA Health and a link to vaccine.gov (where people can find local pharmacies that carry the bivalent booster).
  Arms: Consistency and uniqueness information reminder; Consistency reminder; Eligibility information reminder; Severity information reminder; Simple reminder; Uniqueness information reminder
Behavioral: Consistency framing — The message will leverage the psychological principle of consistency. It will highlight to patients that based on medical records, they have completed a COVID-19 vaccine primary series, have done a great job protecting their health, and can now get the bivalent booster.
  Arms: Consistency and uniqueness information reminder; Consistency reminder
Behavioral: Information provision about the uniqueness of the bivalent booster — The message will contain information about how the bivalent booster differs from previous doses patients have received and why it is valuable.
  Arms: Consistency and uniqueness information reminder; Uniqueness information reminder
Behavioral: Information provision about bivalent booster eligibility — The message will clarify to patients that regardless of whether they are at high risk, received the original boosters, or previously got COVID-19, they are eligible for the bivalent booster based on their medical records, and the updated booster will be valuable for them.
  Arms: Eligibility information reminder
Behavioral: Information provision about the severity of COVID-19 symptoms — The message will contain information about the often underestimated chances of people developing severe or long-lasting COVID-19 symptoms. The message will also mention that the bivalent booster can reduce such chances.
  Arms: Severity information reminder

SUMMARY:
This study investigates different ways to elevate intentions to get the COVID-19 booster via text-based reminders, including providing information about the booster and leveraging the consistency principle. The proposed randomized controlled trial will examine the impact of these reminders on booster uptake.

DETAILED DESCRIPTION:
The proposed randomized controlled trial will take place a few weeks after UCLA Health notified its patients about bivalent COVID-19 boosters. The trial will test whether text-based reminders can increase uptake of bivalent COVID-19 boosters and examine different ways to elevate intentions to get the booster. This trial will include a randomly selected ~40% of patients from all UCLA Health patients eligible to receive the COVID-19 bivalent booster at the time of the study, with 35% of the remaining eligible patients randomly allocated to another trial (Pre-registration title: "Boost intentions and Facilitate Action to Promote Covid-19 Booster Take-up") and 25% randomly allocated to a third trial (Pre-registration title: "Effects of Prompt to Bundle Covid-19 Booster and Flu Shot"). The three trials will be run simultaneously.

Patients randomly selected for this trial will be randomized at an equal share to 7 conditions: an Holdout condition that does not receive a text reminder and 6 additional conditions that receive a text message (simple reminder, uniqueness information reminder, eligibility information reminder, severity information reminder, consistency reminder, and consistency and uniqueness information reminder; see description in the Arm/Interventions section). Within each arm, patients are further randomized into one of the 33 time slots for when they will receive the text message (i.e., 3 time points per day including 9am, 12pm, 4pm for 11 days). Days 1-4 and 8-11 have slightly fewer patients than Days 5-7.

First, to test whether the text reminders increase vaccine uptake, the investigators will compare the holdout condition to the combination of the 6 reminder arms.

The investigators will also investigate additional questions:

1. The investigators will investigate how the information provision strategies affect vaccine uptake. For this purpose, the investigators will compare vaccine uptake and link click rates between (1) the uniqueness information reminder, (2) the eligibility information reminder, and (3) the severity information reminder. If there are significant differences across three information provision reminders in a given outcome, the investigators will separately compare these three reminders with the simple reminder and the holdout arm. If there are not significant differences across the three information provision reminders in a given outcome, the investigators will compare the average of these three reminders with the simple reminder and holdout. The investigators will also compare the simple reminder with the holdout arm. For the severity information reminder, the investigators have competing predictions. On one hand, highlighting underestimated severity may increase the perceived importance of the vaccine; on the other hand, the negative valence of this message may create reactance, leading people to avoid thinking about COVID-19 and vaccination.
2. The investigators will investigate how the consistency framing affects vaccine uptake and whether the combination of consistency and uniqueness information has a positive effect. On one hand, the psychological literature about the consistency principle suggests that people strive to behave consistently with their past actions and positions; thus, reminding people that they have completed the primary series and have done a good job at protecting their health may motivate them to consistently take care of themselves by getting the bivalent booster. On the other hand, patients may get complacent after being reminded that they have already finished the primary series, thinking that they have already completed the necessary steps to protect themselves. Hence, the investigators have competing predictions about whether the consistency framing can effectively increase vaccine uptake. The combination of consistency and uniqueness information about how the bivalent booster differs from the previous doses may be most powerful. To understand the role of consistency framing, the investigators will compare the consistency reminder with the simple reminder (in both vaccine uptake and link click rates) and the holdout condition (in vaccine uptake only). To test the effect of consistency framing and uniqueness information, the investigators will compare the consistency and uniqueness information reminder with the consistency reminder, the uniqueness information reminder, simple reminder, and holdout, respectively.
3. The investigators will explore the role of the time when a text message is sent. The investigators will examine how the effect of text reminders (i.e., the combination of the 6 reminder arms vs. holdout) varies across days and times. As additional specifications, the investigators will control for the time trend and analyze all patients who have not gotten the bivalent booster in California or scheduled a booster appointment at UCLA Health the day before the trial starts.

Analysis:

The investigators will run ordinary least squares regressions (OLS) with robust standard errors to predict the aforementioned outcome variables, except that the investigators will use a Cox proportional hazards model with administrative censoring to predict time of obtaining the booster. The significance level will be 0.05. The regressions will include the following control variables:

* Indicators for one of the 33 time slots
* Participant age (If there will be a missing value, the investigators will replace with the mean and add a dummy variable to indicate patients with missing age)
* Indicators for participant race/ethnicity (Black non-Hispanic, Hispanic, Asian non-Hispanic, white non-Hispanic, other/mixed, unknown)
* Indicators for participant gender (male, female, other/unknown)

The investigators will test whether the main effect of sending text reminders (i.e., the combination of the 6 reminder arms vs. holdout) is robust regardless of:

* Whether the patient is female or male
* Whether the patient is white non-hispanic or racial/ethnical minority
* Whether the patient is 65+ (including 65) or below 65

The investigators will investigate the following moderators for (1) the effect of sending a text reminder to facilitate action and (2) the effect of boosting intentions via information provision; since the investigators have competing predictions about the effectiveness of consistency framing, the investigators will exclude the arms containing consistency framing from this analysis:

* Timing of the first dose of the COVID-19 vaccine primary series
* Whether patients got at least one original booster before the trial starts
* Whether or not the patient received a flu shot in either the 2020-2021 season or the 2021-2022 flu season according to the patient's medical record
* How strongly the patient's neighborhood is in favor of the Republican (vs. Democratic) Party if UCLA Health eventually agrees to provide de-identified addresses (e.g., zip code) and if the sample includes patients living in Republican-leaning counties.

Additional information: Three days into this trial, the investigators learned that the supply of boosters at UCLA Health is very limited and patients could not find appointments at UCLA Health. The investigators verified that local pharmacies continue to have appointments available. Thus, the investigators updated all text messages to (1) explain that UCLA Health has limited booster appointments available, (2) no longer provide a direct link to schedule appointments at UCLA Health, and (3) instead encourage patients to make an appointment at local pharmacies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above
* Have a mobile phone number or SMS-capable phone number in UCLA Health's database
* Having completed a COVID-19 vaccine primary series based on CAIR data
* Last COVID-19 vaccine shot (including booster shot) occurred at least two months before the date when patient list are pulled in preparation for the trial, based on CAIR data. The last two criteria meant to identify patients who are eligible for the updated booster.

Exclusion Criteria:

* Patients who have received the bivalent booster anywhere (based on CAIR data) before the day they receive the text message
* Patients who have already scheduled appointments at UCLA Health for getting the bivalent booster before the day they receive the text message

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177720 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
booster take-up in 2 weeks | 2 weeks after getting the text message
  Whether people receive the bivalent booster at any location reporting to the California Immunization Registry (CAIR)
booster take-up in 4 weeks | 4 weeks after getting the text message
  Whether people receive the bivalent booster at any location reporting to the California Immunization Registry (CAIR)

SECONDARY OUTCOMES:
Link click rate in 1 week | 1 week after getting the text message
  Whether people click on at least one link provided in the text message

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No